CLINICAL TRIAL: NCT02918227
Title: Exploration of Ejaculation Changing Mechanism After Surgery for Benign Prostatic Hyperplasia
Acronym: EMMECH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough patient
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: I15028 (EMMECH)
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Prostate; Ejaculation; Benign Prostatic Hyperplasia
Keywords: Ejaculation; Benign Prostatic Hyperplasia; Prostate
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Search retrograde ejaculation (Experimental): Sperm count (spz) after orgasm achieved by masturbation will be measured, corresponding to the sum of spz collected in the ejaculate (E) and the first urine after orgasm (U). These measures will be made before surgery (E1 and U1) and after surgery (E2 and U2). The values E1, E2, U1 and U2 will be achieved by multiplying the concentration of spz per unit volume by the total volume of collection.
  Interventions: Procedure: Search retrograde ejaculation

INTERVENTIONS:
Procedure: Search retrograde ejaculation — Sperm count (spz) after orgasm achieved by masturbation will be measured, corresponding to the sum of spz collected in the ejaculate (E) and the first urine after orgasm (U). These measures will be made before surgery (E1 and U1) and after surgery (E2 and U2). The values E1, E2, U1 and U2 will be achieved by multiplying the concentration of spz per unit volume by the total volume of collection.

SUMMARY:
Every year in France, more than 60 000 people are operated for benign prostatic hyperplasia (BPH). This surgery is accompanied by a change or even a loss of ejaculations externalized what constitutes the main constraint for patients. Empirically, the investigators talk to the patient "retrograde ejaculation" to explain a possible loss of ejaculation. Yet the underlying mechanism of this modification or loss of ejaculation remains completely unknown. Yet the underlying mechanism of this modification or loss of ejaculation remains completely unknown. No study could not determine whether the predominant mechanism was a real retrograde ejaculation or aspermia. Moreover, technical changes are sometimes tempted to preserve antegrade ejaculation but no scientific rationale can not validate.

DETAILED DESCRIPTION:
Every year in France, more than 60 000 people are operated for benign prostatic hyperplasia (BPH). This surgery is accompanied by a change or even a loss of ejaculations externalized what constitutes the main constraint for patients. Empirically, the investigators talk to the patient "retrograde ejaculation" to explain a possible loss of ejaculation. Yet the underlying mechanism of this modification or loss of ejaculation remains completely unknown. No study could not determine whether the predominant mechanism was a real retrograde ejaculation or aspermia. Moreover, technical changes are sometimes tempted to preserve antegrade ejaculation but no scientific rationale can not validate.

ELIGIBILITY:
Inclusion Criteria:

* Man, at least 18 years, which is scheduled for a BPH surgery
* Sexually active
* Measurement of Residual postvoid less than 6 months
* Patients accepting the constraints of the study
* Signed Consent
* Affiliate or beneficiary of social security system.

Exclusion Criteria:

* Patients unable to understand the study or to give consent
* Patients with known infertility
* Patients previously operated prostate
* Patients previously treated with a natural prostate treatment (radiotherapy, microwave, radio frequency, ultrasound)
* Patients with known urethral stenosis before surgery
* Patient with impaired preoperative in ejaculation
* Patient under guardianship or under judicial protection
* Patient subject to psychiatric care

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-06-11 (Actual)

PRIMARY OUTCOMES:
Sperm count | Baseline and 9 months
  Sperm count (spz) after orgasm achieved by masturbation will be measured, corresponding to the sum of spz collected in the ejaculate (E) and the first urine after orgasm (U). These measures will be made before surgery (E1 and U1) and after surgery (E2 and U2). The values E1, E2, U1 and U2 will be achieved by multiplying the concentration of spz per unit volume by the total volume of collection.
aspermia (A) | Baseline and 9 months
  Aspermia is determined by the ratio of the difference of total spz between before surgery and after surgery on the number of spz before surgery
retrograde ejaculation (R) | Baseline and 9 months
  retrograde ejaculation is determined by the difference in percentage of retrograde ejaculation between postoperative and preoperative
Evaluation of the coefficient C | 9 months
  A and R will be subtracted to obtain the coefficient C

SECONDARY OUTCOMES:
Type of surgery | 9 months
  determination of factors influencing the ejaculation changing mechanism after BPH surgery by evaluation of the coefficient C depending of type of surgery
Preoperative prostate volume | 9 months
  determination of factors influencing the ejaculation changing mechanism after BPH surgery by preoperative prostate volume measurement by ultrasound
Evaluation of the coefficient C depending on changing sexual symptoms relating to the change of sexuality questionary (IIEF15) before and after surgery | Baseline and 9 months
  determination of factors influencing the ejaculation changing mechanism after BPH surgery by changing sexual symptoms relating to the change of sexuality questionary (IIEF15) before and after surgery
Changing in urinary output before and after surgery | Baseline and 9 months
  determination of factors influencing the ejaculation changing mechanism after BPH surgery by changing in urinary output before and after surgery
Evaluation of urinary symptoms questionary (IPSS) before and after surgery | Baseline and 9 months
  determination of factors influencing the ejaculation changing mechanism after BPH surgery by changing in urinary symptoms corresponding to the change in score in the evaluation of urinary symptoms questionary (IPSS) before and after surgery
Degree of resection evaluated by pre/postoperative prostate volume ratio, ratio of prostatic specific antigen (PSA) preoperative / postoperative and measurement of the resected weight (or the number of joules used in case of laser vaporization). | Baseline and 9 months
  determination of factors influencing the ejaculation changing mechanism after BPH surgery by assessment of degree of resection

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien DESCAZEAUD, MD, Principal Investigator — Limoges Univerity Hospital
Locations (3):
- France (3):
  - CHU de LIMOGES, Limoges
  - CHU de Nîmes, Nîmes
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No